CLINICAL TRIAL: NCT05732350
Title: Real-world Exploratory Evaluation of the Potential Drug-drug Interaction Between Anticancer Small Molecule Inhibitors and Direct Oral Anticoagulants in Patients With Solid Tumours and Exploration of the Role of Therapeutic Drug Monitoring
Brief Title: Exploratory Drug Interaction Study Between SMIs and DOACs
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL78003.068.21
Record Dates: First submitted 2023-01-27; First posted 2023-02-17 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor; Cancer, Lung
Keywords: direct oral anticoagulant; targeted therapy; small molecule inhibitors; Therapeutic drug monitoring
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Citrate whole blood samples, EDTA whole blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients in group 1 already receive a DOAC and will start treatement with an SMI. Blood samples will be drawn before start of the SMI and during concomittant use with the SMI.
- Group 2: Patients in group 2 already use a potentially relevant DOAC-SMI combination or already use an SMI and start with a DOAC. In this group, blood samples are taken after the start of concomittant use of the DOAC-SMI combination.

SUMMARY:
The main objective of this study is to investigate the effect of small molecule inhibitors (SMIs), used in targeted therapy for tumours, on direct oral anticoagulants (DOACs).

DETAILED DESCRIPTION:
Patients who receive anticoagulant therapy in the form of a direct oral anticoagulant (DOAC) and simultaneously receive anti-cancer targeted therapy with a small molecule inhibitor (SMI), potentially have an increased risk on thromboembolic complications and bleeding events due to interfering drug-drug interactions. Some SMIs influence CYP3A4 and/or p-glycoprotein (p-gp) for which DOACs are substrates. In this study, the effect of theoretically relevant SMIs on the pharmacokinetics, efficacy and safety of DOACs in patients with solid tumours will be investigated. For this purpose, plasma concentration analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a solid tumour
* 18 years of age or older
* Patients receive or start treatment with an SMI-DOAC combination, that may cause a clinically significant DDI at the level of CYP3A4 and/or P-gp, based on the SmPC
* Combined use of a DOAC-SMI combination is expected to be continued at the same dose for at least three weeks
* The DOAC is used for at least seven days and the SMI has already been used for at least 21 days at time of blood collection to ensure steady-state
* Patients receive a DOAC at maintenance dose

Exclusion Criteria:

* Unable to understand the information in the patient information letter
* Any concurrent medication beside the SMI and DOAC that is known to strongly inhibit or induce CYP3A4 or P-gp
* Patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer who will be, or are already, treated with an SMI and a DOAC simultaneously, at the MUMC+ or Radboudumc can participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
DOAC trough concentration | At least 7 days after start DOAC use and in combination with an SMI at steady-state (after at least 21 days)
  DOAC trough concentration before and during concomitant use with an SMI
DOAC peak concentration | At least 7 days after start DOAC use and in combination with an SMI at steady-state (after at least 21 days)
  DOAC peak concentration before and during concomitant use with an SMI

SECONDARY OUTCOMES:
Thromboembolic and bleeding events during follow-up | within 6 months after the last blood sampling
  Thromboembolic and bleeding events during follow-up
SMI trough concentration during concomitant use with a DOAC | After the start of the DOAC use in combination with an SMI at steady-state (after at least 21 days)
  SMI steady-state trough concentration during concomintant use with a DOAC

OTHER OUTCOMES:
Thrombin generation before and during concomitant use of a DOAC and an SMI | At least 7 days after start DOAC use and in combination with an SMI at steady-state (after at least 21 days)
  Thrombin generation before and during concomitant use of a DOAC and an SMI

CONTACTS AND LOCATIONS:
Overall Officials: Robin van Geel, PharMD, PhD, Principal Investigator — Maastricht UMC
Locations (2):
- Netherlands (2):
  - Radboud UMC, Nijmegen, Gelderland
  - Maastricht UMC, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: No